CLINICAL TRIAL: NCT04881305
Title: Characterizing Long-term Cognitive and Emotional Impairment in Post-COVID-19 Sequelae
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RMC-0939-20
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Post-COVID / Long-COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Adults recovered from COVID-19 (diagnosed using RT-PCR), 3-8 months after the onset of the acute stage of the disease, with cognitive/emotional complaints.
  Interventions: Diagnostic Test: questionnaires and neuropsychological assessment
- Controls: Adults recovered from COVID-19 (diagnosed using RT-PCR), 3-8 months after the onset of the acute stage of the disease, reporting no cognitive/emotional complaints.
  Interventions: Diagnostic Test: questionnaires and neuropsychological assessment

INTERVENTIONS:
Diagnostic Test: questionnaires and neuropsychological assessment — Participants will undergo: (1) An evaluation of COVID-19-related symptoms such as fatigue, post-exertional malaise, dizziness, etc. (2) A comprehensive evaluation of behavioral measures (e.g., hearing, vision, olfaction, sleep, social engagement) (3) A short validated neuropsychological evaluation, of multiple cognitive domains, with an emphasis on the memory domain; motivational factors will also be taken into account using performance validity tests (4) A thorough well-being and emotional state assessment, including the evaluation of mood disturbance and quality of life. The assessment will involve both self-report and cognitive tasks, previously associated with psychopathology. In addition to the above-mentioned evaluations, a subgroup of participants will undergo either MRI examination or FDG PET-CT, with the aim of clarifying the neural mechanisms underlying the neurologically-related symptoms.

SUMMARY:
Weeks and months after they have seemingly recovered from COVID-19, many patients continue to suffer from major long-term effects. While the virus typically hits the respiratory system, accumulating evidence now indicates a variety of other, non-respiratory symptoms, some of which manifest long after recovery from the acute phase of the disease. Neurologically-related symptoms among COVID-19 convalescents include extreme fatigue, headaches, sleep and mood disorders, cognitive decline and long-lasting impairments in the gustatory and olfactory systems. Interestingly, it seems that there is no direct link between the severity of the disease in its acute stage and the existence or the severity of the long-lasting symptoms. This means that to date, the possibility that even patients who present mild to moderate symptoms will still go on to develop long-lasting neuropsychiatric disorders following the disease cannot be ruled out. Unfortunately, most of the scientific literature relies on self-report of recovered patients and on qualitative assessments of healthcare workers. The literature still lacks a quantified objective characterization of these long-term impairments. Such data ought to be collected using designated questionnaires and validated neuropsychological assessments.

In order to allow for a better understanding of the biological mechanisms that underlie long-term effects of COVID-19, comprehensive research in this population is required. Alongside the identification of the variety of symptoms involved, the importance of an interdisciplinary approach that will take into account the emotional and cognitive aspects of the patients is necessary. Patients need accurate information about the possible consequences of this disease, in order to reduce their anxiety and, if needed, to allow them and their family members and caretakers to prepare for the comings. A systematic characterization of the mental effects of COVID-19 will allow global healthcare systems to develop prevention and rehabilitation programs and provide psychological and/or psychiatric follow-up and intervention programs, according to circumstances. By elucidating the mechanisms underlying emotional and cognitive deficits in COVID-19 convalescents, this study may improve future management of the consequences of the pandemic, potentially contributing to the development of efficient medical treatments for populations who suffer from the long-term effects of the disease.

DETAILED DESCRIPTION:
70 participants (above 18 years of age) will be recruited from the post-COVID recovery clinic at the Beilinson Hospital, in the Rabin Medical Center (RMC). Only patients previously diagnosed using reverse transcription-polymerase chain reaction (RT-PCR), and that had no neurological or psychiatric disease prior to the COVID-19 episode, will be included. To avoid the risk of measuring adverse effects of lack of oxygen and/or artificial respiration procedures, COVID-19 patients who suffered from severe acute disease (according to World Health Organization criteria) will be excluded from participation. All potential participants will be given a detailed explanation about the research goals and procedure and they will all be asked to sign an institutional review board (IRB) consent form. Two groups, matched for age (5± years), will be examined: 35 case study patients: convalescents who report suffering from cognitive/emotional decline after recovering from COVID-19, and 35 control cases: convalescents with no cognitive/emotional complaints Participants will undergo: (1) An evaluation of COVID-19-related symptoms such as fatigue, post-exertional malaise, dizziness, etc. (2) A comprehensive evaluation of behavioral measures (e.g., hearing, vision, olfaction, sleep, social engagement) (3) A short validated neuropsychological evaluation, of multiple cognitive domains, with an emphasis on the memory domain; motivational factors will also be taken into account using performance validity tests (4) A thorough well-being and emotional state assessment, including the evaluation of mood disturbance and quality of life. The assessment will involve both self-report and cognitive tasks, previously associated with psychopathology. By recruiting a heterogeneous cohort in terms of symptom severity, the investigators will be able to test possible correlations between the emotional and cognitive impairments. In addition to the above-mentioned evaluations, a subgroup of participants will undergo either magnetic resonance imaging (MRI) or fluorodeoxyglucose (FDG)-positron emission tomography (PET)-computed tomography (CT), with the aim of clarifying the neural mechanisms underlying the neurologically-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic individuals who recovered from COVID-19, 3-8 months after the onset of the acute stage of the disease. All individuals will be Israeli citizens, fluent Hebrew speakers with normal/corrected to normal vision and hearing abilities.

Exclusion Criteria:

* Asymptomatic convalescents, and symptomatic convalescents who have a history of one or more of the following: Chronic obstructive pulmonary disease (COPD), Congestive heart failure (CHF), ischemic heart disease (IHD), Cerebrovascular accident (CVA), Chronic Kidney disease (CKD) with glomerular filtration rate of less than 30ml/minute, Cirrhosis of the liver, Hypoxia (less than 80% oxygen levels at room air), neurologic disease, diagnosed decline in cognitive function prior to disease onset , psychiatric disease or usage of anti-psychotic medications, addiction to drugs or alcohol.

In addition, a potential participant will be excluded from participation if he/she has a contraindication to magnetic resonance (MR) scanning, as defined by the Rabin Medical Center regulations: this includes patients with unremovable non-MR compatible implants, pregnant women and participants who suffer from claustrophobia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
cognitive/emotional impairment | at time of testing (3 - 8 months after diagnosis)
  abnormal outcome in the neuropsychological assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel